CLINICAL TRIAL: NCT05319691
Title: Yoga for Chronic Low Back Pain: A Type 1 Hybrid Implementation-Effectiveness Pragmatic Randomized Control Trial in the Cleveland Clinic Employee Health Plan
Brief Title: Yoga for Chronic Low Back Pain in the Cleveland Clinic Employee Health Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Saper (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Robert Saper, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-132
Record Dates: First submitted 2022-02-04; First posted 2022-04-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain; Back Pain
MeSH Terms: conditions — Chronic Pain; Back Pain | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Investigators will use a single-blinded (investigator) two-arm randomized control trial (RCT) design. The trial will be 24 weeks long and divided into two distinct parts: an initial 12-week Treatment Phase followed by a 12-week Follow-up Phase. Participants will be randomized 1:1 into weekly virtual yoga classes (Yoga Now) or a wait-list control (Yoga Later) who will receive usual care. After the 24 week study period, participants in Yoga Later will be offered the yoga intervention in a non-study format.
Who Masked: Investigator
Masking Description: Investigators will use a single-blinded (investigator) two-arm randomized control trial (RCT) design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Now (Treatment Group) (Active Comparator): An initial 12-week Treatment Phase of weekly virtual yoga classes (Yoga Now) followed by a 12-week Follow-up Phase.
  Interventions: Behavioral: Yoga
- Yoga Later (Wait List Control Group) (No Intervention): A wait-list control group (Yoga Later) will receive usual care. After the 24 week study period, participants in Yoga Later will be offered the yoga intervention in a non-study format.

INTERVENTIONS:
Behavioral: Yoga — The trial will be 24 weeks long and divided into two distinct parts: an initial 12-week Treatment Phase during which, yoga participants will receive a reproducible standardized weekly yoga intervention delivered virtually with additional resources for home practice, followed by a 12-week Follow-up Phase.
  Other Names: Treatment Group; Yoga Now
  Arms: Yoga Now (Treatment Group)

SUMMARY:
This study uses clinical trial and implementation science methodology to specifically assess the effectiveness of yoga into the management of chronic low back pain (cLBP) within the Cleveland Clinic Employee Health Plan. The study will use a type 1 hybrid effectiveness-implementation design, which tests a clinical intervention while collecting data on implementation. Studying and implementing evidence-based, non-pharmacologic interventions is an important strategy for improving pain management and reducing opioid use disorder.

DETAILED DESCRIPTION:
The investigators will use a single (investigators) blinded two-arm randomized control trial (RCT) design. The trial will be 24 weeks long and divided into two distinct parts: an initial 12-week Treatment Phase followed by a 12-week Follow-up Phase. Participants will be randomized 1:1 into weekly virtual yoga classes (Yoga Now group) or a wait-list control (Yoga Later group) who will receive usual care. After the 24 week study period, participants in the Yoga Later Group will be offered the yoga intervention in a non-study format as well as a free yoga mat and access to online yoga for LBP videos.

The screening and enrollment process will all occur remotely and involves the following: 1) A telephone or Information Technology approved, The Health Insurance Portability and Accountability Act (HIPAA-secure), virtual meeting platform where participants provide consent for completion of eligibility screening through a standardized questionnaire; 2) if eligible, provision of information about the study presented by study personnel with use of an Institutional Review Board approved information page for informed consent, answering all questions about the study, and assuring participant understanding through the "teach back" method.

Randomization occurs after administering the baseline survey. Investigators will use a computerized randomization procedure built into the study management system, RedCap, to randomize each enrolled participant using a 1:1 ratio to the Yoga Now group or Yoga Later group. Permuted variably-sized block randomization with block sizes of 6, 12 and 18 will be used.

The study interventions start within approximately one week of baseline data collection and randomization. Participants will be asked to complete questionnaire forms at baseline, weeks 6, 12 and 24. All participants throughout the entire 24-week study can continue to receive routine medical care including doctor visits and pain medication.

The hatha yoga intervention, a term for yoga that pairs poses and breathing techniques, is structured and reproducible. The full instructor manual and participant manual are available online. Originally, it was developed by an expert panel led by Rob Saper, MD and Master of Public Health (MPH) in 2007 and used in a pilot study of 30 participants with cLBP. It was further refined in 2011 in a dosing study of 95 participants and a larger non-inferiority trial of 320. It is designed specifically for the yoga-naïve individual for effectiveness and safety in cLBP. Each class is 75 minutes long and will be delivered virtually to a maximum class size of 12. Yoga instructors will complete an 8-hour training on the protocol directed by the Cleveland Clinic lead yoga instructor.

Class begins with a relaxation exercise, yoga breathing exercises, and a brief discussion of yoga philosophy. The class proceeds with warm-up yoga exercises and then yoga postures. Yoga breathing is emphasized throughout. The class ends with a relaxation exercise. The 12 weeks are divided into four 3-week segments. Each segment is given a theme (e.g., "Listening to the Wisdom of the Body"). Participants are frequently advised to go slowly and carefully. The degree of difficulty of postures learned increases with each segment. For each segment, the participants gradually learn a sequence of 12-15 poses. The protocol provides variations and uses various aids (e.g., chair, strap) to accommodate a range of physical abilities. Participants are strongly encouraged to practice at home for 30 minutes daily on days which they do not attend yoga class. To facilitate home practice, participants will be given a free yoga mat, participant manual, and provided access to online videos prepared by the study instructors.

Ten percent of online yoga classes will be virtually observed and assessed by a study team member for instructor fidelity to the protocol using a checklist. A 12-week follow-up phase consisting of larger optional classes for maintenance will follow.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* Current non-specific LBP persisting ≥12 weeks with average pain intensity ≥4 for the previous week on an 11-point numerical rating scale
* Ability to speak and understand English

Exclusion Criteria:

* Any severe psychiatric or medical comorbidity in the Principal Investigator's judgment that would make study participation unsafe or not feasible.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Self-reported average pain intensity for the previous week | Baseline
  11 point numerical rating scale ranging from 0=no pain to 10=worst possible pain
Change of self-reported average pain intensity for the previous week | Week 12
  11 point numerical rating scale ranging from 0=no pain to 10=worst possible pain
Self-reported back-related function | Baseline
  Modified Roland Morris Disability Questionnaire ranging from 0=no functional impairment to 23=worst impairment of function
Change of self-reported back-related function | Week 12
  Modified Roland Morris Disability Questionnaire ranging from 0=no functional impairment to 23=worst impairment of function

SECONDARY OUTCOMES:
Change of self-reported average pain intensity for the previous week | Week 24
  11 point numerical rating scale ranging from 0=no pain to 10=worst possible pain
Change of self-reported back-related function | Week 24
  Modified Roland Morris Disability Questionnaire ranging from 0=no functional impairment to 23=worst impairment of function
Analgesic use | Baseline
  Self-reported pain medications usage; dosage reported in milligrams
Analgesic use | Week 12
  Change of self-reported pain medications usage; dosage reported in milligrams
Analgesic use | Week 24
  Change of self-reported pain medications usage; dosage reported in milligrams
Global improvement | Weeks 12 and 24
  Overall improvement by self-report (6-point Likert scale, 1 = very worse to 6 = very improved).
Patient Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 - Pain Interference - Short Form 4a | Weeks 12 and 24
  PROMIS Pain domain asks 4 questions. Each question is rated from 1 to 5. Values are summed to create a total raw score. Raw scores are minimum 4 to maximum 20 and translate to a T score with a minimum 41.6 to maximum 75.6. A higher score equates to a higher pain interference.

OTHER OUTCOMES:
Total Medical Expenditures for low back pain | Baseline to Week 24
  Total and back-related medical expenditures for all participants for the six month study period will be compared between the yoga (Arm 1) and wait-list (Arm 2) control groups.
  Cost of implementing the intervention will be measured to demonstrate the feasibility of evaluating cost-effectiveness of yoga compared to usual care for cLBP from the perspective of the payer.
Participant Satisfaction | Baseline to week 24
  Acceptability will be measured by participant satisfaction with treatment (5-point Likert scale, 1 = very dissatisfied to 5 = very satisfied) and answers to open-ended questions about the effect of yoga, facilitators and barriers.
Sleep Quality | Baseline to week 24
  Overall change in sleep quality from baseline to weeks 6, 12 and 24, measured by PROMIS Sleep disturbance Short Form 8a, item #1, range: 0-4, with higher scores reflecting better sleep quality. Raw score at each time point will used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Saper, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Saper RB, Sherman KJ, Delitto A, Herman PM, Stevans J, Paris R, Keosaian JE, Cerrada CJ, Lemaster CM, Faulkner C, Breuer M, Weinberg J. Yoga vs. physical therapy vs. education for chronic low back pain in predominantly minority populations: study protocol for a randomized controlled trial. Trials. 2014 Feb 26;15:67. doi: 10.1186/1745-6215-15-67. PMID 24568299
- [Background] Saper RB, Sherman KJ, Cullum-Dugan D, Davis RB, Phillips RS, Culpepper L. Yoga for chronic low back pain in a predominantly minority population: a pilot randomized controlled trial. Altern Ther Health Med. 2009 Nov-Dec;15(6):18-27. PMID 19943573
- [Background] Saper RB, Boah AR, Keosaian J, Cerrada C, Weinberg J, Sherman KJ. Comparing Once- versus Twice-Weekly Yoga Classes for Chronic Low Back Pain in Predominantly Low Income Minorities: A Randomized Dosing Trial. Evid Based Complement Alternat Med. 2013;2013:658030. doi: 10.1155/2013/658030. Epub 2013 Jun 26. PMID 23878604
- [Background] Saper RB, Lemaster C, Delitto A, Sherman KJ, Herman PM, Sadikova E, Stevans J, Keosaian JE, Cerrada CJ, Femia AL, Roseen EJ, Gardiner P, Gergen Barnett K, Faulkner C, Weinberg J. Yoga, Physical Therapy, or Education for Chronic Low Back Pain: A Randomized Noninferiority Trial. Ann Intern Med. 2017 Jul 18;167(2):85-94. doi: 10.7326/M16-2579. Epub 2017 Jun 20. PMID 28631003
- [Derived] Tankha H, Gaskins D, Shallcross A, Rothberg M, Hu B, Guo N, Roseen EJ, Dombrowski S, Bar J, Warren R, Wilgus H, Tate P, Goldfarb J, Drago VG, Saper R. Effectiveness of Virtual Yoga for Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2442339. doi: 10.1001/jamanetworkopen.2024.42339. PMID 39485352